CLINICAL TRIAL: NCT02742272
Title: Development of a Clinical Decision Rule to Identify Pediatric Patients With Headache at Low Risk for Intra-cranial Pathology
Brief Title: Clinical Decision Rule for Pediatric Intracranial Pathology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1506-076
Record Dates: First submitted 2015-11-20; First posted 2016-04-19 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Migraine Headache; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ED Headache or Migraine Patients: The investigators will perform a prospective cohort study of patients ages 6-18 years presenting to the ED with a complaint of headache or migraine over a 12 month period.

SUMMARY:
The purpose of this study is to develop a clinical decision rule for patients seen in the pediatric emergency department for possible intracranial pathology. This a prospective study evaluating patients presenting with headache and migraine. The study is observational and does not impact patient care.

DETAILED DESCRIPTION:
Background/Question: A significant number of children who present to the Emergency Department (ED) with headache or migraine undergo head imaging with Computed Tomography (CT) or Magnetic Resonance Imaging (MRI). However, there is relatively low yield in imaging neurologically normal patients based on prior studies. The goal of this study is to describe the utilization of head CT or MRI among pediatric ED patients with headache and migraine. The investigators plan to evaluate clinical and examination characteristics of these patients, and use this information to develop a clinical decision rule to help providers predict the risk of finding an abnormality that affects patient treatment.

Design: The investigators will perform a study of all children between 6 and 18 years of age who present to the ED with headache or migraine. At the time of the visit providers will be asked to complete a questionnaire regarding exam and history without making any changes to patient care. The investigators will also contact a sub-group of patients who do not undergo MRI or CT, 12-14 weeks after discharge to ask about subsequent headache care after leaving our facility.

Methods: All children age 6-18 years who present to the ED with a chief complaint of headache or migraine will be eligible for the study. Patients will be excluded if they meet any of the following criteria: trauma within 48 hours, previous neurosurgery (shunt included), known tumor, history of cerebral hemorrhage/ischemia, Sickle Cell Disease, thrombophilia, bleeding disorder or non-English speaker. ED Research Assistants and ED staff physicians and nurse practitioners will screen potential candidates and ask providers to review the inclusion criteria. If the eligibility criteria are met, the provider will complete a standardized data collection form regarding exam and history findings. Patient care will not be impacted or altered. Research Assistants will also provide a Parent Information Sheet (either during the visit, or by mail following the ED visit) to the family of those patients who are enrolled informing them they may be contacted following discharge. Medical records will be reviewed for all eligible patients to obtain information on patient demographics, course of treatment and diagnosis. For those patients who do not have any head CT or MRI performed at their visit, the family will be contacted 12-14 weeks later to determine if they have had subsequent care for their headache. If the family is unable to be reached by phone, the patient chart will be reviewed for any other pertinent visits.

Analysis: For each patient characteristic examined, the investigators will look for a statistically significant difference between those patients who have normal head imaging, and those with abnormal imaging. Using the characteristics that are significantly different, the investigators will develop a clinical decision rule to help providers assess the risk of significant findings in an individual patient. The investigators will also develop a decision tree to help aid providers when deciding which patients need head imaging. A sample of patients will have two independent assessments to allow us to look for evidence of inter-rater reliability in our questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years
* Chief complaint of headache or migraine

Exclusion Criteria:

* Exclusion criteria
* Head trauma within 48 hours
* Previous neurosurgery (shunt included)
* Personal history of brain tumor
* History of stroke or vascular abnormality
* Sickle Cell Disease
* Fever (temperature over 38 degrees C)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients presenting to the ED with Headache or Migraine who meet the inclusion criteria and do not meet any exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Intracranial pathology identified by imaging studies | within 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Cain, MD, Principal Investigator — Children's Minnesota
Locations (1):
- Children's Hopsitals and Clinics of Minnesota, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larson DB, Johnson LW, Schnell BM, Goske MJ, Salisbury SR, Forman HP. Rising use of CT in child visits to the emergency department in the United States, 1995-2008. Radiology. 2011 Jun;259(3):793-801. doi: 10.1148/radiol.11101939. Epub 2011 Apr 5. PMID 21467249